CLINICAL TRIAL: NCT04006561
Title: Prospective Neurobehavioral Evaluation in Newly-diagnosed Patients With Primary CNS Lymphoma Treated With Hyperfractionated Conformal Whole-brain Radiation Therapy Plus Simultaneous Integrated Boost
Brief Title: Prospective Neurobehavioral Functions in Newly-diagnosed Patients With Primary CNS Lymphoma Treated With Hyperfractionated Conformal Whole-brain Radiation Therapy Plus Simultaneous Integrated Boost
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1812140031
Record Dates: First submitted 2019-06-18; First posted 2019-07-05 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-03

CONDITIONS: Primary CNS Lymphoma; Brain Lymphoma
Keywords: Primary CNS Lymphoma; Neurobehavioral Assessment; Neurocognitive Function (NCF); Whole-Brain Radiation Therapy (WBRT); Simultaneous Integrated Boost (SIB); Hyperfractionation; Radiotherapy; Chemotherapy; Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly-diagnosed patients with primary CNS lymphoma
  Interventions: Radiation: A treatment protocol of combined chemoradiation delivered in the manner of hyperfractionated conformal whole-brain radiation therapy

INTERVENTIONS:
Radiation: A treatment protocol of combined chemoradiation delivered in the manner of hyperfractionated conformal whole-brain radiation therapy — Each freshly-diagnosed patient with primary CNS lymphoma will be treated with combined chemoradiation in a sandwiched way, in which 2 cycles of induction chemotherapy with intravenous methotrexate (MTX in a conventional dose of 1g/m2) and intrathecal MTX are followed by a complete course of hyperfractionated WBRT and then high-dose cytarabine for 2 cycles.

SUMMARY:
Primary central nervous system lymphoma (PCNSL) is an uncommon disease. Conventional treatment has consisted of either whole-brain radiation therapy (WBRT) or methotrexate (MTX)-based combined modality therapy integrating chemotherapy with cranial irradiation in a sandwiched manner. No matter whether the dosage of MTX is high or conventional, combining chemotherapy with WBRT greatly improves intracranial tumor control and even survival outcomes. However, delayed treatment-related neurotoxicity and neurocognitive sequelae emerged as a significant debilitating complication in PCNSL patients, especially when effective combined chemoradiation can achieve disease control and long-term survival rates. Therefore, by delivering hyperfractionated conformal WBRT plus SIB, this prospective cohort study aims to accomplish both optimal intracranial control and minimal WBRT induced neurocognitive decline. Additionally, by administering objective multi-domain neurobehavioral/neurocognitive assessments, the change in neurocognitive functions (NCFs) before and after the course of hyperfractionated conformal WBRT will be investigated and analyzed.

According to the treatment guidelines for treating newly-diagnosed PCNSL patients, combined chemoradiation in which the WBRT course is sandwiched between initial courses of MTX and the later courses of chemotherapy with Ara-C is the treatment of mainstay at our institute. Employing the technique of a conformal CT treatment planning, the WBRT course is delivered in the manner of hyperfractionation with a reduced cumulative dose of 3600 cGy in 30 fractions during 3-4 weeks, administered twice daily in 1.2 Gy - fractions with at least 6 hours between fractions. By virtue of multidisciplinary management and teamwork including neurosurgery, hematology, radiation oncology, and neuroimaging expertise, it is attempted to recruit all potentially eligible patients with newly-diagnosed PCNSL. Most importantly, a professional neuropsychologist participates in this research project to integrate neurobehavioral outcomes into the prospective study. Accordingly, a battery of neuropsychological measures is used to evaluate predetermined NCFs for the studied patients. The test battery is composed of six standardized neuropsychological tests, covering four domains sensitive to disease and treatment effects (executive function, attention, verbal memory, information processing). The primary outcome measure is the change in patients' capability of information processing indicated by the Paced Auditory Serial Addition Test-Revised (PASAT-R), from the baseline before receiving the WBRT course to the follow-up after undergoing the entire courses of combined chemoradiation.

This prospective cohort study aims to thoroughly examine newly diagnosed PCNSL patients by using a standard battery of neurobehavioral/neurocognitive functions. Additionally, a better intracranial disease control is expected since the WBRT course relies on a highly conformal treatment planning integrated with the individualized arrangement of simultaneous integrated boost (SIB) to escalate the focal dose irradiating the originally involved site(s). Moreover, WBRT-related neurocognitive sequelae might be significantly less likely to occur because the WBRT course is delivered in the fashion of hyperfractionation, indicating a significantly lower dose per fraction and a reduced cumulative dose. Furthermore, it is anticipated the investigators will analyze which neurobehavioral domain would predict the treatment-related neurocognitive impacts to the largest extent in newly diagnosed PCNSL patients treated with cranial RT combined with or without MTX based chemotherapy according to the multidisciplinary treatment guidelines implemented at a single institute.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histopathologic diagnosis of non-Hodgkin's lymphoma (NHL) by brain biopsy
* A typical MRI/CT scan for primary CNS lymphoma is defined as the presence of hypo, iso, or hyperintense parenchymal contrast-enhancing (usually homogeneously) mass lesion(s)
* Patients must have a normal or negative pre-treatment systemic evaluation including: i. A bone marrow aspirate and biopsy ii. CT scans of the chest, abdomen and pelvis iii. Patients must have adequate bone marrow reserve
* Patients must be HIV-1 negative
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment

Exclusion Criteria:

* A past history of major psychiatric disease
* Prior cranial irradiation for any reasons
* Other active primary cancer with the exception of basal cell carcinoma of skin and cervical carcinoma in situ
* Pre-existing immunodeficiency such as renal transplant recipient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly-diagnosed patients with primary CNS lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2029-02-18 (Estimated); Study Completion 2029-02-18 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the change in patients' capability of information processing, as determined by the assessment (the Paced Auditory Serial Addition Test-Revised) from baseline up to 30 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 30 months after completing all courses of chemoradiation
  The Paced Auditory Serial Addition Test-Revised is an assessment of information processing, used to assess the capacity and speed of information processing, as well as sustained and divided attention.
The primary endpoint is delayed recall, as determined by the change/decline in verbal memory (Word Sequence Learning Test) from baseline up to 30 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 30 months after completing all courses of chemoradiation
  The Word Sequence Learning Test is an assessment of verbal memory. To evaluate auditory memory of verbal information without context.
The primary endpoint is the change of executive function, as determined by three different domains assessments from baseline up to 30 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 30 months after completing all courses of chemoradiation
  The Modified Card Sorting Test is an assessment of executive function, related to conceptual formation and mental shifting.
The primary endpoint is the change of executive function, as determined by three different domains assessments from baseline up to 30 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 30 months after completing all courses of chemoradiation
  The Trail Making Test is an assessment of speed and flexibility, used to measure the ability of visual attention and task switching.
The primary endpoint is the change of executive function, as determined by three different domains assessments from baseline up to 30 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 30 months after completing all courses of chemoradiation
  The Semantic Association of Verbal Fluency Test is an assessment of verbal fluency, related to frontal and temporal cortex.
  A measure of the ability of phonemic and semantic variants.
The change in attention functions from baseline up to 30 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 30 months after completing all courses of chemoradiation
  Neurocognitive assessment including: Paced Auditory Serial Addition Test-Revised

SECONDARY OUTCOMES:
The time from the date of recruitment to that of intracranial progression/failure noted on brain MRI | Baseline before the WBRT course; 2 months after completing all courses of chemoradiation, and follow up to 30 months
Depression Inventory questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and follow up to 30 months
  Questionnaires include: Beck Depression Inventory (BDI). The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, used psychometric tests for measuring the severity of depression.
  The BDI contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Anxiety Inventory questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and follow up to 30 months
  Questionnaires include: Beck Anxiety Inventory (BAI). The Beck Anxiety Inventory (BAI) is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.
  The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are:
  0-7: minimal anxiety; 8-15: mild anxiety; 16-25: moderate anxiety; 26-63: severe anxiety.
Self & family Evaluation questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and follow up to 30 months
  Questionnaires include: National Taiwan University Irritability Scale Self Evaluation(NTUIS-Self), National Taiwan University Irritability Scale-Family Evaluation (NTUIS-Family).
  The National Taiwan University Irritability Scale (NTUIS) is a self-reported scale with validated and reliable psychometric properties, to specifically evaluate irritability.
  The NTUIS required patients to examine their irritability before and after disease.
  The NTUIS is a 6-point Likert scale with 18 items. Each item was rated 1 (totally non-matched to patient's conditions) to 6 (totally matched to patient's conditions) with descriptions anchoring each matching level. Since "excessive emotional (e.g. anger and annoyance) and behavioural (e.g. verbal aggression) responses to stimuli" were used as the operational definition of irritability, the items considering anger, verbal aggression and annoyance were selected.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan